CLINICAL TRIAL: NCT04944459
Title: Meditation Utilizing Signals From Electroencephalography in Chronic Pain (MUSE-PAIN) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center For Interventional Pain and Spine (Other)
Collaborators: InteraXon (Unknown); Celéri Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MUSE-PAIN
Record Dates: First submitted 2021-06-01; First posted 2021-06-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muse-S (Experimental): multi-sensor neurofeedback-assisted mindfulness training device (Muse-S)
  Interventions: Device: Muse-S headband; InteraXon Inc., RRID:SCR_014418

INTERVENTIONS:
Device: Muse-S headband; InteraXon Inc., RRID:SCR_014418 — Muse-S is used as a technology-supported Mindfulness Training (tsMT) device as a way to introduce meditation as a method for managing chronic pain in individuals as it facilitates the learning process, requires minimal training to use and provides mechanisms to enhance compliance and track progress. The availability of direct feedback data from Muse-S may encourage the participant to perform meditation sessions and may increase time spent in the "calm" brain state.

SUMMARY:
This clinical investigation is a prospective, open-label, non-randomized, multi-center study. It is designed to assess the use of the Muse-S meditation system in patients with chronic pain based on clinical follow-up data and exploratory cold pressor testing.

Baseline assessments will be taken prior to exposure to Muse-S. Subjects will be followed for 7 weeks for main study endpoints and will continue to be followed through 12 months during a study extension period.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, open-label, non-randomized, multi-center study. It is designed to collect clinical follow-up data on the use of the Muse-S headband system in patients with chronic pain.

Adult chronic pain patients without systematic meditation experience will be eligible to participate in this study.

After signing the informed consent form (ICF), patients will enter the screening/baseline period. Screening/baseline assessments will include data collection (including previous Electronic Medical Record (EMR) data), patient self-reported questionnaires and cold pressor testing.

Subjects will receive and be trained on the Muse-S headband system and will be asked to perform daily assigned intervention with the Muse device for 7 weeks during the main study period, which will include at a minimum achieving 2 new chapters per week in the pain course until the pain course is completed, a minimum of Muse mind sessions 3 times per week at a minimum of 5 minutes per session and engagement with the Muse system at a minimum of 5 times per week once the pain course is complete. Patients will be instructed to do Muse Mind Meditation on the Muse App for a minimum of 5 minutes daily and will be required to complete the entire pain course content during the main study period. Functional device data will be collected during all Muse sessions. In addition, study participants have the option to use the Muse-S go to sleep journey and to sleep with the device if they are comfortable doing so in order in order to provide data on their sleep sessions.

During this main study period, investigative sites will follow up with study participants after baseline to answer any study-related questions and assess for any device-related AEs, which will include two follow up telephone calls at day 3 (± 1 day) and week 4 (± 3 day) to assess patient satisfaction and their ability to use the device. In addition, subjects will be required to respond remotely to patient self-reported questionnaires on a weekly basis.

The main study portion for a study participant will end when the final main study visit is completed [7 weeks post start of study intervention (±1 week)], which will include cold pressor testing.

Following completion of the main study, subjects will be encouraged to continue using their Muse-S device for the next 12 months during a study extension period. During this extension period, functional device data will be collected following all Muse-S sessions with patient self-reported questionnaires and EMR data collection at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to provide written informed consent prior to any clinical study-related procedure.
2. Subject is at least 18 years (or the minimum age required by local law to consent for participation in a clinical investigation) or older at the time of enrollment.
3. Subject has had a chronic painful condition for more than 3 months.
4. Subject is on stable background treatment for at least 6 weeks prior to starting Muse therapy (i.e., no changes to any medical device(s) used or pharmaceutical agents administered for pain, mood, sleep or spasm, including change to dose or interval).
5. Subject is naïve to the regular practice of any form of meditation.
6. Subject has access to the following personal devices with regular internet access for completion of study-related assessments and interventions:

   * Access to an iPhone, iPad or Android capable device and/or computer for the purposes of electronically completing patient self-reported questionnaires via SMS text or email.
   * Access to an iPhone or iPad (i.e., an Apple device) in order to interact with the Muse-S Headband system, the Muse App and the Meditation Studio App. Refer to the following link for details regarding which Apple devices are compatible with Muse: https://choosemuse.force.com/s/article/What-devices-are-compatible-with-Muse?language=en_US. (NOTE: Meditation Studio App, which is used for the pain course, can only accommodate Apple devices. Therefore, only Subjects with access to an Apple device can initially be enrolled. However, there are future plans to also have the pain course available on the Muse App. Once the pain course is available on the Muse App, the Meditation Studio App will no longer be needed and Subjects with Android devices will also be eligible for participation at that time.)
7. Subject has medical clearance to perform activities that somebody of their age and level of physical fitness could reasonably do without doing irreparable damage to their body (i.e., patient will not be harmed if they resume normal activity upon alleviation of any of their pain).
8. Subject, in the opinion of the Investigator, is able to understand this clinical investigation, cooperate with the investigational procedures, operate the Muse-S device, and is willing to complete remote assessments and return for follow-up.

Exclusion Criteria:

1. Subject is enrolled, or intends to participate, in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug, or additional testing beyond standard of care procedures) which could confound the results of this trial as determined by the investigator (e.g., another clinical or research program which intervenes on the patient's pain, stress, anxiety or Quality of Life).
2. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements (e.g., cognitive deficits, history of head injury or a neuropsychological or psychiatric condition or use of psychoactive drugs that may influence the functioning of the central nervous system).
3. Any condition that would preclude the subject from participating in cold pressor testing based on the investigator's opinion such as history of Raynaud's phenomena, syncope, cardiovascular disorder, or frostbite or has an open cut, sore, or bone fracture on or near their hand to be submersed.
4. Subject frequently engages in cold therapy (practice of using cold water or ice baths to treat health conditions or stimulate health benefits (also known as cold hydrotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Changes in PROMIS-29 scores relative to baseline. | Baseline, 7 weeks, 6- and 12 months
  Changes from PROMIS-29 scores relative to baseline for each domain evaluated (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity). The first seven domains are assessed with 4 questions each; Pain Intensity is measured with a single 11-point numeric rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain). High scores represent more of the domain being measured. Thus, on symptom-oriented (negatively-worded) domains of PROMIS-29 (anxiety, depression, fatigue, pain interference, and sleep disturbance), higher scores represent worse symptomatology. On the function-oriented (positively-worded) domains (physical functioning and social role) higher scores represent better functioning.
Change in Pain Impact Score (PIS) (calculated from PROMIS-29) relative to baseline. | Baseline, 7 weeks, 6- and 12 months
  The Pain Impact Score (PIS) is a derivative of the PROMIS-29 that ranges from 8 (low impact) to 50 (high impact). The PIS is calculated by adding the raw scores for pain intensity [0-10] and pain interference [4-20] along with the inverted raw score for physical function [4-20].
Change in Patient Global Impression of Change (PGIC) relative to baseline. | 7 weeks, 6- and 12 months
  Subjects will be asked if their overall pain was very much improved, much improved, minimally improved, no change, minimally worse, much worse or very much worse.

SECONDARY OUTCOMES:
Change in Numeric Rating Scale (NRS) by pain area(s) relative to baseline. | Baseline, 7 weeks, 6- and 12 months
  Patients will be asked to rate their pain area(s) using a 0 to 10 numeric rating scale (NRS). 0 being no pain and 10 being the worst pain imaginable.
Percent Pain Relief (PPR) by pain area(s) relative to baseline. | 7 weeks, 6- and 12 months
  Patients will be asked on a scale of 0-100, with 100% being complete relief and 0% being no relief, how much relief from their pain area(s).
Impact of study intervention on Pain Catastrophizing by assessing change in Pain Catastrophizing Scale (PCS) relative to baseline. | Baseline, 7 weeks, 6- and 12 months
  The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking (degree to which people experience an aversive orientation towards pain) according to 3 components: rumination, magnification, and helplessness. It consists of 13 items rated on a 0-4 scale, with a total range of 0 to 52. Respondents will rate the frequency in which they experience such thoughts on a scale ranging from 0 (not at all) to 4 (all the time). A lower score indicates a better result.
Patient Engagement | 7 weeks
  Adherence to Muse use by summarizing the frequency of use.
Patient Satisfaction | 7 weeks, 6-, and 12-months
  Patients will be asked a series of Patient Satisfaction and Engagement Questions where they will respond to questions using a five point Likert Scale (Strongly Agree; Agree; Neutral; Disagree; Strongly Disagree).

OTHER OUTCOMES:
Changes in Heart Rate Variability (HRV) during and after cold pressor test (acute phase), and after completion of protocol (chronic phase) | Baseline and 7 weeks
Changes in Peak Alpha Frequency during and after cold pressor test (acute phase), and after completion of protocol (chronic phase) | Baseline and 7 weeks
Changes in cold pressor test time in seconds during cold pressor test (acute phase), and after completion of protocol (chronic phase) | Baseline and 7 weeks
  Cold pain threshold - time to the first report of pain and cold pain tolerance - time to removal of the hand from the ice bath (measured in seconds postsubmersion).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fishman, MD, Principal Investigator — Center For Interventional Pain and Spine
Locations (2):
- United States (2):
  - Pacific Research Institute, LLC, Santa Rosa, California
  - Center For Interventional Pain and Spine, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center For Interventional Pain and Spine — https://centerpain.com/